CLINICAL TRIAL: NCT01470417
Title: GAIN-1 Study: Gemcitabine With Abraxane and Other Investigational Therapies in Neoadjuvant Treatment of Pancreatic Adenocarcinoma
Brief Title: Gemcitabine With Abraxane and Other Investigational Therapies in Neoadjuvant Treatment of Pancreatic Adenocarcinoma
Acronym: GAIN-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701386; GAIN-1 (Other: University of Florida)
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Albumin-Bound Paclitaxel; Gemcitabine; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): Individuals with low risk disease will receive nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with low risk disease will have an additional two cycles of therapy (4 total cycles) prior to resection.
  Interventions: Drug: Chemotherapy
- Chemotherapy and ChemoRadiotherapy (Active Comparator): Individuals with high-risk disease or borderline resectable disease will receive nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with high-risk or borderline resectable disease will receive additional chemotherapy with radiation therapy prior to resection.
  Interventions: Drug: Chemotherapy + ChemoRadiotherapy

INTERVENTIONS:
Drug: Chemotherapy — Nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with low risk disease will have an additional two cycles of therapy (4 total cycles) prior to resection.
  Other Names: Abraxane; Gemcitabine
  Arms: Chemotherapy
Drug: Chemotherapy + ChemoRadiotherapy — Nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with high-risk or borderline resectable disease will receive additional chemotherapy with radiation therapy prior to resection.
  Other Names: Abraxane; Gemcitabine
  Arms: Chemotherapy and ChemoRadiotherapy

SUMMARY:
This study will evaluate the role of Gemcitabine and Abraxane in the treatment of resectable and borderline-resectable pancreatic cancer by giving the chemotherapy before surgery.

DETAILED DESCRIPTION:
This current study proposes to conduct a prospective non-randomized open-label phase II trial using Gemcitabine and Abraxane in the neoadjuvant treatment of resectable and borderline-resectable pancreatic cancer. For patients that are low-risk resectable (based on prediction rule) the plan is to administer 2 cycles of Gemcitabine and Abraxane followed by additional systemic therapy or chemotherapy with radiation therapy (chemoRT), followed by surgical resection. For patients who are either borderline-resectable or high-risk resectable (see schema), the plan is to administer 2 cycles of Gemcitabine and Abraxane followed by chemoradiotherapy concurrent with gemcitabine followed by surgical resection. For those without high-risk features, systemic chemotherapy alone will be administered. The primary endpoints will be R0 surgical resection rate, biochemical (CA 19-9), pathologic and radiologic response rates. Secondary endpoints will include progression-free survival (PFS), overall survival (OS), 30-day post-op mortality, toxicity, quality of life, pain control, and correlative molecular exploratory analysis involving pancreatic tumor and stromal SPARC expression levels. The investigators will also assess the patient, tumor, and clinical characteristics that may predict R0 resectability, thus further refining the predictive rule in high-risk patients as defined by Bao and colleagues. The investigators' hypothesis is that by using targeted and risk-adapted chemotherapy or chemoRT, improved R0 surgical resections can be achieved and effective systemic therapy delivered, which will translate to a significant improvement in overall survival in patients with pancreatic adenocarcinoma, compared to published historical controls.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically or cytologically confirmed adenocarcinoma of the pancreas.

  * Patients must have locally advanced pancreatic cancer, classified as either low-risk resectable (LR), high-risk resectable (HR) or borderline resectable (BR)
  * Age between 18 and 90 years at the time of consent.
  * Patients with biliary obstruction must have adequate drainage prior to starting treatment.
  * Patients must have ≤ Grade I peripheral neuropathy (CTCAE v 4.0)
  * Patients must have ≤ ECOG Performance status 2
  * Pretreatment laboratory parameters:

    * Absolute granulocyte/neutrophil count (AGC/ANC) ≥ 1.8 thou/mm3
    * Platelet count ≥ 100,000/mm3
    * Bilirubin < 2 mg/dl
    * ALT/SGPT < 10x upper limit of normal
    * Creatinine < 3 mg/dl
    * Calculated creatinine clearance (via Cockcroft-Gault) > 30 mL/min
    * Baseline CA 19-9 levels
  * Signed study specific, IRB stamped informed consent

Exclusion Criteria:

* • Evidence of any distant metastasis including peritoneal seeding and/or malignant ascites

  * Previous irradiation to the abdomen that would compromise the ability to deliver the prescribed treatment
  * Prior treatment for pancreatic cancer
  * Active, untreated infection
  * Surgical resection of the tumor (not including biopsies)
  * Other malignancy (except non-melanoma skin cancer) that has not been disease-free for at least 5 years.
  * Pregnant and/or breast-feeding women, or patients (men and women) of child-producing potential not willing to use medically acceptable contraception while on treatment and for at least 3 months thereafter.
  * Use of anti-epileptics (drugs such as phenytoin, phenobarbitol and carbamazepine)
  * ECG abnormality with the following: QTC >500, left bundle branch block or any other clinically significant finding that would interfere with protocol therapy.
  * History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas George, MD, FACP, Principal Investigator — University of Florida
Locations (1):
- University of Florida Shands Cancer Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy + ChemoRadiotherapy: Individuals with high-risk disease or borderline resectable disease will receive nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with high-risk or borderline resectable disease will receive additional chemotherapy with radiation therapy prior to resection.
  Chemotherapy and ChemoRadiotherapy: Nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with high-risk or borderline resectable disease will receive additional chemotherapy with radiation therapy prior to resection.
Period: Overall Study
Arm/Group | Chemotherapy | Chemotherapy + ChemoRadiotherapy
Started | 3 | 7
Completed | 3 | 5
Not Completed | 0 | 2
Not completed — Disease progression | 0 | 2

BASELINE CHARACTERISTICS:
Population: Adults with pathologically confirmed resectable or borderline resectable pancreatic adenocarcinoma
Groups:
- Chemotherapy + ChemoRadiotherapy: Individuals with high-risk disease or borderline resectable disease will receive nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with high-risk or borderline resectable disease will receive additional chemotherapy with radiation therapy prior to resection.
  Chemotherapy + ChemoRadiotherapy: Nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with high-risk or borderline resectable disease will receive additional chemotherapy with radiation therapy prior to resection.
- Total: Total of all reporting groups
Arm/Group | Chemotherapy | Chemotherapy + ChemoRadiotherapy | Total
Number analyzed (Participants) | 3 | 7 | 10
Age, Continuous [Mean (Full Range); unit: years] | 69.3 [64 to 78] | 67.3 [55 to 78] | 67.9 [55 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Response Rate
Description: Biochemical response rate (serum CA 19-9). Baseline compared to pre-operative serum CA19-9 values.
Time Frame: 4 - 8 weeks after neoadjuvant therapy
Population: The seven subjects included in this analysis had CA19-9 testing performed at baseline and again prior to surgery. Pre-operative CA19-9 testing was not performed for one subject so they were not included in this analysis nor were two subjects who were found to have progressive disease prior to completing neoadjuvant therapy.
Measure: Mean (Full Range); unit: U/mL
Arm/Group | Chemotherapy | Chemotherapy + ChemoRadiotherapy
Number analyzed (Participants) | 3 | 4
U/mL
  Baseline CA19-9 | 383 [2 to 1036] | 550 [1 to 1833]
  Pre-Operative CA19-9 | 43 [1 to 109] | 53 [1 to 141]

2. Primary Outcome: Radiographic Response Rate
Description: Evaluate radiographic response of the measurable disease with repeat imaging at 4 - 8 weeks after therapy. Measurable disease was evaluated using Response Evaluation Criteria In Solid Tumors Criteria (RECIST) 1.1 criteria. Per RECIST v1.1 in target lesions assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), >20% growth in the sum of the longest diameter or target lesions or appearance of new lesions; Stable Disease (SD), change in sum of longest diameter of target lesions does not meet criteria for PR or PD. The number of subjects experiencing Complete Response (CR), Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD) is reported.
Time Frame: 4 - 8 weeks after neoadjuvant therapy
Population: All subjects enrolled in the study were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Chemotherapy | Chemotherapy + ChemoRadiotherapy
Number analyzed (Participants) | 3 | 7
participants
  Partial Response | 1 | 0
  Stable Disease | 2 | 5
  Progressive Disease | 0 | 2

3. Primary Outcome: Pathologic Downstaging and Margin Status
Description: Pathologic stage and margin status after resection. Pathologic downstaging was determined my looking at the rate of R0 (all residual tumor removed during surgery) vs R1 (microscopic tumor present at the resection margin per pathology) resections.
Time Frame: At the time of surgery after neoadjuvant therapy
Population: Subjects who had a surgical resection of their primary tumor were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Chemotherapy | Chemotherapy + ChemoRadiotherapy
Number analyzed (Participants) | 3 | 5
participants
  R0 Resection | 3 | 3
  R1 Resection | 0 | 2

4. Secondary Outcome: 90 Day Post-operative Mortality
Description: Evaluate mortality in the first 90 days after surgery
Time Frame: 90 days after surgery
Measure: Number; unit: participants
Arm/Group | Chemotherapy | Chemotherapy + ChemoRadiotherapy
Number analyzed (Participants) | 3 | 5
participants
  Number of survival | 3 | 5
  Number of mortality | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from informed consent to 30 days following the last dose of protocol therapy.
Groups:
- Chemotherapy and ChemoRadiotherapy: Individuals with high-risk disease or borderline resectable disease will receive nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with high-risk or borderline resectable disease will receive additional chemotherapy with radiation therapy prior to resection.
  Chemotherapy and ChemoRadiotherapy: Nab-paclitaxel 100 mg/m2 IV over 30 minutes on days 1, 8, and 15 along with gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 in an every 28 day cycle for two cycles. Subjects with high-risk or borderline resectable disease will receive additional chemotherapy with radiation therapy prior to resection.
Arm/Group | Chemotherapy | Chemotherapy and ChemoRadiotherapy
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/7
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=3) | Chemotherapy and ChemoRadiotherapy (N=7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=3) | Chemotherapy and ChemoRadiotherapy (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Alopeica (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (4) | 5 (8)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dsgeusia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (Gastrointestinal disorders) | 3 (8) | 6 (17)
Fever (General disorders) | 0 (0) | 2 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (7) | 2 (6)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Investigations) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (4) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nervous system disorders - Other, autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (5)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 3 (5)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes